CLINICAL TRIAL: NCT04593238
Title: Effect of Double Antibiotic Paste Versus Calcium Hydroxide as Intra-canal Medications on RANKL/OPG Levels and Periapical Bone Healing in Patients With Asymptomatic Apical Periodontitis: A Randomized Clinical Trial
Brief Title: Effect of Double Antibiotic Paste Versus Calcium Hydroxide on RANKL/OPG Levels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Amr Saad Mohamed Elsayed, Assitant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDO: 3-3-6
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Biological Markers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Double antibiotic paste intra-canal medication group (n=25) (Experimental): 500 mg Metronidazole tablet+ 500 mg Ciprofloxacin tablet crushed into powder and mixed together with salline to form a creamy mix to be placed inside the root canal for 1 week.
  Interventions: Drug: Double Antibiotic paste
- Calcium hydroxide intra-canal medication group (n=25) (Active Comparator): Calcium hydroxide paste (Metapaste) placed inside the root canal for 1 week
  Interventions: Drug: Calcium Hydroxide Paste - Non-Setting

INTERVENTIONS:
Drug: Double Antibiotic paste — Metronidazole and Ciprofloxacin
  Other Names: Bimix
  Arms: Double antibiotic paste intra-canal medication group (n=25)
Drug: Calcium Hydroxide Paste - Non-Setting — Calcium hydroxide paste to be delivered inside the canal as an intra-canal medication
  Other Names: Metapaste
  Arms: Calcium hydroxide intra-canal medication group (n=25)

SUMMARY:
The aim of the present study is to evaluate the effect of double antibiotic paste when compared to Ca (OH)2, in terms of RANKL and OPG levels in chronic periapical lesions and correlate the results with periapical bone healing findings after a follow up period of one year.

DETAILED DESCRIPTION:
Apical periodontitis is an inflammatory disease that occurs as a consequence of the bacterial infection of dental pulp tissue. It represents an inflammatory/immune pathogenesis affecting the periapical tissue including the surrounding bone. This periapical process is primarily initiated by bacterial infection in the necrotic pulp. Its persistence, progression to chronic lesions and destruction of bone structures are a consequence of the inability of host-defense mechanisms to eradicate infection. Periapical lesions are characterized histologically by fibrous and granulated tissue, infiltrated by different inflammatory cells.

Up to now the diagnosis and follow-up of asymptomatic apical periodontitis AAP is based on a clinical radiographic evaluation, however, this reflects the accumulated damage from previous episodes of periodontal tissue destruction. Moreover, the clinical presentation does not reflect the underlying inflammatory response. In accordance, differences in disease severity involve qualitatively and quantitatively different inflammatory responses. Nowadays, the challenge focuses on the necessity of designing innovative non-invasive chair-side point-of-care assessment methods, accounting for the biological profile as a complement to the existing clinical-radiographic assessment to contribute to the early evaluation of treatment outcome.

Rationale for conducting the research:

When dental pulp is infected or inflamed, various inflammatory mediators, including cytokines, chemokines, and neuropeptides, are released by innate and adaptive immune cells. During the development of pulp inflammation, inflammatory mediators result in the formation of apical osteolytic lesions. Bone loss is mainly caused by activated osteoclasts. Various cytokines such as interleukin (IL)-1, IL-11, IL-17, and tumor necrosis factor alpha (TNF-a) stimulate osteoclast progenitor cell differentiation and activation by the osteoprotegerin (OPG)/nuclear factor kappa B ligand (RANKL)/nuclear factor kappa B (RANK) complex.

The molecular mechanisms underlying bone resorption are regulated by the interaction between RANKL and OPG.The interaction between RANKL and RANK is necessary for the differentiation and activation of osteoclasts. This is modulated by OPG, which, in turn, suppresses osteoclast differentiation by preventing the interaction between RANKL and RANK.The production of OPG and RANKL by different cell types is regulated by local and systemic stimuli, including bacterial products, hormones, and inflammatory mediators.Changes in the balance of the mediators determine the progression and severity of bone diseases such as those found in periapical and periodontal lesions.

It has been reported that antibiotics regulate the immune response through modulation of cytokines production. Therefore, the level of cytokines, RANKL, and OPG can also be affected by antibiotics. In the infected root canal system, virulence products, antigens, and microbial cells are the main causes of apical periodontitis. Microorganisms in the root canal system adhere to root canal walls, isthmuses, ledges and commonly formed biofilm communities.The application of antimicrobial intra-canal medication is recommended to eliminate bacteria that could not be removed from the root canal system after instrumentation and irrigation of the root canals.

Calcium hydroxide (Ca (OH)2) is generally preferred in endodontics as an intracanal medicament because of its antimicrobial and biological effects. Because of its solubility, Ca (OH)2 releases calcium and hydroxyl ions slowly providing an alkaline environment in the periapical region.

There has been only a single in vivo study performed to evaluate the effect of Ca (OH)2 combined with ciprofloxacin or ibuprofen on the release of RANKL/OPG in periapical lesions. The aim of the present study is to evaluate the effect of double antibiotic paste when compared to Ca (OH)2, in terms of RANKL and OPG levels in chronic periapical lesions and correlate the results with periapical bone healing findings after a follow up period of one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are free from any physical or mental handicapping conditions and with no underlying systemic diseases.
* Age between 20-45years old.
* Males & Females.
* Single canaled teeth:

  * Diagnosed clinically with asymptomatic apical periodontitis.
  * Absence of spontaneous pain
  * Size of periapical radiolucency: 2-4 mm (i.e. score 3 according to CBCT periapical index proposed by Estrela)30, including only the tested tooth.
* Patients who didn't use any NSAIDs or antibiotics for 1 month before treatment.
* Patients' acceptance to participate in the trial.

Exclusion Criteria:

* - Medically compromised patients.
* Pregnant women.
* Patients reporting bruxism or clenching.
* Patients allergic to ciprofloxacin or metronidazole.
* Teeth associated with acute periapical abscess and/or swelling.
* Greater than grade I mobility or pocket depth greater than 5mm.
* Size of periapical radiolucency is less than 2 mm or greater than 4 mm.
* Non restorable teeth.
* Immature teeth.
* Radiographic evidence of external or internal root resorption vertical root fracture, perforation, calcification.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Percentage change of RANKL/OPG levels | measured Immediately post-instrumentation and after one week
  RANKL/OPG levels will be measured post-instrumentation and 1 week postoperatively, using Absorbance using ELISA test, to calculate the percentage change of RANKL/OPG levels

SECONDARY OUTCOMES:
Periapical healing | CBCT scans will be done preoperatively and 6 and 12 months postoperatively
  Periapical healing will be evaluated using CBCT (The lesion size is given a score according to the CBCT periapical index proposed by Estrela